CLINICAL TRIAL: NCT07286422
Title: Efficacy of Subclavian Vein/Artery Diameter Index in Predicting the Incidence of the Spinal-Induced Hypotension in Geriatric Patients: A Prospective, Observational Study.
Brief Title: Efficacy of Subclavian Vein/Artery Diameter Index in Predicting the Incidence of the Spinal-Induced Hypotension in Geriatric Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, tarek abdel hay mostafa, principle investigator, Tanta University
Other Study IDs: SCV with hypotension
Record Dates: First submitted 2025-12-02; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Spinal Induced Hypotension; Old Age; Debility
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Assessment of the SCV & SCA — The right SCV was measured using a linear array probe, placed in the sagittal plane at the deltopectoral triangle (beneath the proximal part of the middle of the clavicle and the area below the clavicle). In M-mode, measurements of SCV internal anteroposterior diameter, which is maximum during expiration (SCVmax) and minimum during inspiration (SCVmin), were taken in one respiratory cycle.
  Ultrasound scan of the patient's supraclavicular area showing the subclavian artery.
  The index was calculated as the ratio between the SCV maximum diameter and the SAD diameter
Diagnostic Test: Assessment of the IVC and aorta — The IVC measurement will be obtained in the M-mode scan using a curvilinear (3.5 to 5 MHz) ultrasound transducer.
  The transducer was placed longitudinally in the subxiphoid region. The IVC maximum and minimum anterior-posterior diameters were obtained just distal to the IVC-hepatic vein junction. In M-mode, measurements of IVC internal anteroposterior diameter, which is maximum during expiration (IVCmax) and minimum during inspiration. IVCmin), were taken in one respiratory cycle.
  The abdominal aorta was identified to the left of the IVC, 10 mm above the coeliac trunk. The maximum internal anterior-posterior diameter of the aorta was obtained during systole.
  The caval /aorta diameter index was calculated as the ratio between the IVC maximum diameter and the aortic diameter. The index had a sensitivity of 96%, a specificity of 88%, and an accuracy of 95% to predict PSAH at a cut-off point of less than 1.2

SUMMARY:
The hypothesis of the study will be that the subclavian vein/subclavian artery diameter (SCVD/SCAD) index will be a good predictor of spinal-induced hypotension in geriatric patients.

DETAILED DESCRIPTION:
Ultrasonography (USG)-guided measurement of inferior vena cava (IVC) diameters and IVC collapsibility index (IVCCI) are reliable indicators of intravascular volume status and of clinical response to volume resuscitation.

The cava/aorta index had previously shown good ability in assessing volume status and predicting post-spinal hypotension.

The subclavian vein (SCV) is advantageous for measurement as it's supported by the clavicle, preventing deformation or compression. It is also not affected by pregnancy, obesity, or abdominal pain, and its anatomical position remains fixed.

The hypothesis of the study will be that the subclavian vein/subclavian artery diameter (SCVD/SCAD) index will be a good predictor of spinal-induced hypotension in geriatric patients.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients aged 65 or older. 2. Lower body surgeries to be done with spinal anesthesia. 3. BMI less than 30 kg/m2. 4. Patients with ASA I-III.

Exclusion Criteria:

- 1. Patient refusal. 2. Patients with a history of peripheral arterial disease or atherosclerosis 3. Patients with a body mass index of greater than 30 kg/m2 4. Major bloody surgeries (class C surgeries) 5. Patients with a history of cardiovascular disorders, including arrhythmias, heart failure, tricuspid or mitral regurgitation, dilated right atrium or ventricle, AF, ejection fraction < 45%, uncontrolled hypertension, systolic blood pressure <90 mmHg, dyspnea, agitation.

6. Patients with increased intra-abdominal pressure, intra-abdominal mass compressing the IVC.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: 107 geriatric patients, aged 65 or older, scheduled for elective surgery under spinal anesthesia
Sampling Method: Probability Sample
Enrollment: 107 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
subclavian vein to artery index | pre-anesthesia peroid
  The index will be calculated as the ratio between the SCV maximum diameter and the SAD diameter.

CONTACTS AND LOCATIONS:
Locations (1):
- tarek Abdelhay Mostafa, Tanta, El Gharbyia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided